CLINICAL TRIAL: NCT05693727
Title: Cancer Ratio,Pleural Fluid Adenosine Deaminase,Lactate Dehydrogenase, interferonY, Tumor Necrosis Factor,and Interleukins{2,12,18}for Differentiation Between Malignant and Non Malignant Pleural Effusion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mona Adel, Doctor, Assiut University
Other Study IDs: Malignant pleural effusion
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: pleural markers — Pleural Fluid Adenosine Deaminase,Lactate Dehydrogenase, interferonY, Tumor Necrosis Factor,and Interleukins{2,12,18}

SUMMARY:
To evaluate the ability of cancer ratio and pleural fluid markers to discriminate between malignant and non malignant effusion

DETAILED DESCRIPTION:
Pleural effusion is a common clinical entity affecting approximately 1.5 million patients per year in the United States. {3.1}A large number of diseases may be associated with pleural effusion.

This includes:

* Local conditions affecting the pleura (eg, tuberculous pleurisy, pleural mesothelioma),
* Extrapulmonary diseases with secondary pleural involvement (eg, chronic heart failure, liver cirrhosis).

To date, differentiation between both types of pleural effusion (exudate and transudate) is the most common initial diagnostic approach for patients with pleural effusion.

Exudative effusion is commonly seen in three conditions namely cancer (MPE), tuberculosis (TB) and para pneumonic Although MPE can be diagnosed by simple pleural fluid cytology, this method has significant limitations, including a highly variable sensitivity, ranging from as low as 11.6% to as high as 71%.

In contrast to other common causes of pleural effusion such as T.B, no accurate biomarkers of MPE have been established.

Several tumor markers were extensively evaluated, including carcinoembryonic antigen, cytokeratin-19 fragments, and cancer antigen 125, but none of them were found sensitive and specific enough to be implemented in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients (100 cases) with exudative pleural effusion who will be admitted to Department of Chest diseases and Tuberculosis, Assiut University Hospital

Exclusion Criteria:

* Age ˂ 18 years
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with exudative pleural effusion who will be admitted to Department of Chest diseases and Tuberculosis, Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Differentiate between malignant and non malignant pleural effusion by pleural markers | Baseline
  using pleural markers

SECONDARY OUTCOMES:
Time saving | Baseline
  decrease the need for invasive maneuvers for diagnosis
  * decrease length of hospital stay
  * decrease the development of complications

REFERENCES:
- See also: Saguil A, Wyrick K, Hallgren J. Diagnostic approach to pleural effusion. Am Fam Physician. 2014 Jul 15;90(2):99-104. PMID: 25077579. — https://pubmed.ncbi.nlm.nih.gov/25077579/
- See also: Ashutosh Nath Aggarwal, Ritesh Agarwal, Inderpaul Singh Sehgal, Sahajal Dhooria. Adenosine deaminase for diagnosis of tuberculous pleural effusion: A systematic review and meta-analysis. PLoS ONE 14(3): e0213728 — https://pubmed.ncbi.nlm.nih.gov/30913213/